CLINICAL TRIAL: NCT00355927
Title: Changes of the Neuronal Activity in the Subthalamic Nucleus Under Propofol Sedation During Stereotactic Electrode Implantation.
Brief Title: Sedation During Microelectrode Recordings Before Deep Brain Stimulation for Movement Disorders.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DBSsed1-HMO-CTIL; HTA3769
Record Dates: First submitted 2006-07-23; First posted 2006-07-25 (Estimated); Last update posted 2007-11-02 (Estimated); Status verified 2006-08

CONDITIONS: Movement Disorders; Parkinson Disease; Parkinsonian Disorders; Dystonia; Tourette Syndrome
Keywords: Deep brain stimulation; Microelectrode recordings; Basal Ganglia; Sedation; Propofol
MeSH Terms: conditions — Movement Disorders; Parkinson Disease; Parkinsonian Disorders; Dystonia; Tourette Syndrome | interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Sedation with IV propofol — Propofol(50 microgram/kg/min.), I.V. for 5-10 minutes, Until a level of light sedation is achieved
  Other Names: DIPROFOL 1%; TAROPharmceutical Indusries Ltd. IL.

SUMMARY:
The purpose of this study is to detect possible changes in the electrical activity of the Basal Ganglia related to sedation during deep brain stimulation surgery.

DETAILED DESCRIPTION:
Deep Brain Stimulation is commonly used for the treatment of movement disorders. Electrode positioning is usually performed under local anesthesia in fully awake patients. The procedure is uncomfortable to the patients who have to remain motionless during the whole surgery. Previous reports of electrode positioning under general anesthesia was found to be less accurate. This result was probably due to the effect of the anesthetics on the electrical activity of the Basal Ganglia.

The purpose of this study is to detect possible changes in the electrical activity of the Basal Ganglia related to propofol sedation. Electrical activity of single neurons will be recorded before and after sedation.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for Deep Brain Stimulation Surgery.
* Informed concent obtained.

Exclusion Criteria:

* Suspected difficult intubation (by history or physical examination).
* Allergy to Propofol, eggs or soy-beans.
* History of sleep apnea syndrome.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-09; Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
Changes in the electrical activity of neuron cells of the basal ganglia in the examined patients | Within 24 hours needed to analyse the data

CONTACTS AND LOCATIONS:
Overall Officials: Dan Eimerl, MD, Principal Investigator — Hadassah Medical Organization; Zvi Israel, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Israel Z, Hassin-Baer S. Subthalamic stimulation for Parkinson's disease. Isr Med Assoc J. 2005 Jul;7(7):458-63. PMID 16011063
- [Background] Maltete D, Navarro S, Welter ML, Roche S, Bonnet AM, Houeto JL, Mesnage V, Pidoux B, Dormont D, Cornu P, Agid Y. Subthalamic stimulation in Parkinson disease: with or without anesthesia? Arch Neurol. 2004 Mar;61(3):390-2. doi: 10.1001/archneur.61.3.390. PMID 15023817
- [Background] Limousin P, Krack P, Pollak P, Benazzouz A, Ardouin C, Hoffmann D, Benabid AL. Electrical stimulation of the subthalamic nucleus in advanced Parkinson's disease. N Engl J Med. 1998 Oct 15;339(16):1105-11. doi: 10.1056/NEJM199810153391603. PMID 9770557
- [Derived] Benady A, Zadik S, Eimerl D, Heymann S, Bergman H, Israel Z, Raz A. Sedative drugs modulate the neuronal activity in the subthalamic nucleus of parkinsonian patients. Sci Rep. 2020 Sep 3;10(1):14536. doi: 10.1038/s41598-020-71358-3. PMID 32884017
- [Derived] Raz A, Eimerl D, Zaidel A, Bergman H, Israel Z. Propofol decreases neuronal population spiking activity in the subthalamic nucleus of Parkinsonian patients. Anesth Analg. 2010 Nov;111(5):1285-9. doi: 10.1213/ANE.0b013e3181f565f2. Epub 2010 Sep 14. PMID 20841416